CLINICAL TRIAL: NCT05785624
Title: A Two-Cohort, Phase II, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating the Efficacy and Safety of Vixarelimab Compared With Placebo in Patients With Idiopathic Pulmonary Fibrosis and in Patients With Systemic Sclerosis-Associated Interstitial Lung Disease
Brief Title: A Study Evaluating the Efficacy and Safety of Vixarelimab in Participants With Idiopathic Pulmonary Fibrosis and in Participants With Systemic Sclerosis-Associated Interstitial Lung Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to discontinue the study after review of clinical data by the iDMC. This decision was based on unblinded evaluation of clinical efficacy which showed a trend towards futility & was not related to any safety concerns of vixarelimab.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GB44496; 2022-502828-42 (EudraCT Number); 2022-502828-42-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis; Systemic Sclerosis With Lung Involvement
Keywords: Systemic Sclerosis-Associated Interstitial Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- DBT: Cohort 1: Vixarelimab (Experimental): Participants with IPF will receive vixarelimab, subcutaneously (SC), once every two weeks (Q2W) for 52 weeks in the DBT period. This cohort has completed enrollment and has been closed.
  Interventions: Drug: Vixarelimab
- DBT: Cohort 1: Placebo (Placebo Comparator): Participants with IPF will receive vixarelimab matching placebo, SC, Q2W for 52 weeks in the DBT period. This cohort has completed enrollment and has been closed.
  Interventions: Drug: Placebo
- DBT: Cohort 2: Vixarelimab (Experimental): Participants with SSC-ILD will receive vixarelimab, SC, Q2W for 52 weeks in the DBT period.
  Interventions: Drug: Vixarelimab
- DBT: Cohort 2: Placebo (Placebo Comparator): Participants with SSC-ILD will receive vixarelimab matching placebo, SC, Q2W for 52 weeks in the DBT period.
  Interventions: Drug: Placebo
- OLE Period: Cohort 1: Vixarelimab (Experimental): Participants with IPF who complete 52 weeks of treatment in the DBT period can choose to enroll in the OLE period to receive vixarelimab, SC, Q2W for 52 weeks.
  Interventions: Drug: Vixarelimab
- OLE Period: Cohort 2: Vixarelimab (Experimental): Participants with SSC-ILD who complete 52 weeks of treatment in the DBT period can choose to enroll in the OLE period to receive vixarelimab, SC, Q2W for 52 weeks.
  Interventions: Drug: Vixarelimab

INTERVENTIONS:
Drug: Vixarelimab — Vixarelimab will be administered as per the schedule specified in the respective arms.
  Other Names: RO7622888; KPL-716
  Arms: DBT: Cohort 1: Vixarelimab; DBT: Cohort 2: Vixarelimab; OLE Period: Cohort 1: Vixarelimab; OLE Period: Cohort 2: Vixarelimab
Drug: Placebo — Placebo will be administered as per the schedule specified in the respective arms.
  Arms: DBT: Cohort 1: Placebo; DBT: Cohort 2: Placebo

SUMMARY:
The main purpose of the study is to evaluate the efficacy of vixarelimab compared with placebo on lung function in participants with idiopathic pulmonary fibrosis (IPF) and in participants with systemic sclerosis-associated interstitial lung disease (SSc-ILD). Participants who complete 52-weeks of treatment in the Double-blind Treatment (DBT) period can choose to enroll in the optional Open-label Extension (OLE) period to receive treatment with vixarelimab for another 52 weeks.

Cohort 1 has completed enrollment and has been closed for further enrollment. Cohort 2 is enrolling participants.

ELIGIBILITY:
Inclusion Criteria for all Participants:

* FVC ≥45% predicted during screening as determined by the over-reader
* Forced expiratory volume in 1 second (FEV1)/FVC ratio >0.70 during screening as determined by the over-reader
* DLco ≥30% and ≤90% of predicted during screening (Hgb corrected) as determined by the over-reader
* Minimum 6-MWT distance of 150 m with maximum use of 6 liters per minute (L/min) at sea-level and up to 8 L/min at altitude (> 5000 feet [1524 m] above sea level) of supplemental oxygen while maintaining oxygen saturation of >83% during the 6MWT during screening
* Participant and investigator consideration of all medicinal treatment options and/or possibly lung transplantation prior to consideration of participation in the study

Inclusion Criteria for Cohort 1:

* Age 40-85 years
* Documented diagnosis of IPF or IPF (likely)
* HRCT pattern consistent with the diagnosis of IPF, confirmed by central review of chest HRCT and central review of any available lung biopsy
* For participants receiving pirfenidone or nintedanib treatment for IPF: treatment for ≥3 months with a stable dose for ≥4 weeks prior to screening and during screening, with plans to continue treatment during the study period

Inclusion Criteria for Cohort 2:

* Age 18-85 years
* Diagnosis of SSc as defined using the American College of Rheumatology/European Alliance of Associations for Rheumatology (EULAR) criteria
* HRCT demonstrating ≥10% extent of fibrosis, confirmed by central review of Chest HRCT
* Evidence of progression of pulmonary fibrosis
* For participants receiving tocilizumab treatment for SSc-ILD: treatment for ≥3 months with a stable dose for ≥4 weeks prior to screening and during screening, with no contraindications according to local prescribing information, and no intention to change or modify their treatment regimen for the duration of the study
* For participants receiving nintedanib treatment for SSc-ILD: treatment for ≥ 3 months with a stable dose for ≥ 4 weeks prior to screening and during screening, with no contraindications according to local prescribing information, and no intention to change or modify their treatment regimen for the duration of the study
* Availability of skin for biopsy preferably on proximal forearms having Modified Rodnan Skin Score (mRSS) ≥2 at the biopsy location

Inclusion Criteria for OLE Period:

* Completion of 52 weeks of treatment in the double-blinded treatment period
* Investigator determination of a favorable benefit-risk for the individual participant, i.e., the expectation of reasonable likelihood for therapeutic benefit and tolerability of the study drug after evaluation of the preceding 52 weeks of double-blinded treatment

Exclusion Criteria for all Participants:

* Percentage of predicted FVC value showing improvement in the 6-month period prior to screening and including screening value
* Known post-bronchodilator response in FEV1 and/or FVC (defined as an increase in percent predicted values by ≥ 10)
* Resting oxygen saturation of <89% using up to 4 L/min of supplemental oxygen at sea level and up to 6 L/min at altitude (5000 feet [1524 m] above sea level) during screening
* History of lung transplant
* Previous treatment with vixarelimab
* Acute respiratory or systemic bacterial, viral, or fungal infection either during screening or prior to screening not successfully resolved by 4 weeks prior to screening visit
* Presence of pulmonary hypertension requiring treatment
* History of malignancy within the 5 years prior to screening
* Positive hepatitis C virus (HCV) antibody test result accompanied by a positive HCV ribonucleic acid (RNA) test at screening
* Known immunodeficiency
* Known evidence of active or untreated latent tuberculosis

Exclusion Criteria for Cohort 1:

* Evidence of other known causes of ILD
* Emphysema present on ≥50% of the HRCT, or the extent of emphysema is greater than the extent of fibrosis, according to central review of the HRCT

Exclusion Criteria for Cohort 2:

* Evidence of other known causes of ILD
* Rheumatic autoimmune disease other than SSc
* Receiving pirfenidone treatment within 4 weeks prior to screening
* Receipt of nintedanib in combination with tocilizumab

Exclusion Criteria for OLE Period:

* Significant non-compliance in the double-blinded treatment period, per investigator's judgment
* Any new clinically significant pulmonary disease other than IPF or SSc-ILD since enrolling in the double-blinded treatment period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Cohorts 1 and 2: Absolute Change From Baseline in Forced Vital Capacity (FVC) | Baseline up to Week 52
  FVC is a pulmonary function test parameter that indicates the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It's measured by spirometry, which is a common breathing test to check lung function.

SECONDARY OUTCOMES:
Cohorts 1 and 2: Absolute Change From Baseline in 6-Minute Walk Test (6MWT) Distance | Baseline up to Week 52
  The 6MWT test is performed indoors on a flat, straight corridor with a hard surface at least 30 meters (m) in length. 6MWT measures the distance a participant is able to walk quickly on a flat, hard surface in a period of 6 minutes. 6MWT measure will be calculated as the simple difference between baseline distance walked over 6 minutes and week 52 distance walked over 6 minutes as measured in meters.
Cohorts 1 and 2: Absolute Change From Baseline in Percentage of Predicted FVC | Baseline up to Week 52
  FVC is a pulmonary function test parameter that indicates the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It's measured by spirometry, which is a common breathing test to check lung function.
Cohorts 1 and 2: Change From Baseline in Diffusion Capacity of the Lung for Carbon Monoxide Adjusted for Hemoglobin (DLco [Hb]) | Baseline up to Week 52
  DLCO measures the ability of the lungs to transfer gas from inhaled air to the red blood cells in the blood. DLCO is adjusted for hemoglobin as small changes in hemoglobin concentration can affect the carbon monoxide transfer.
Cohorts 1 and 2: Time to Disease Progression | From the start of study treatment until disease progression or death, whichever occurs first (up to Week 52 of DBT)
  Time to disease progression is defined as time to first occurrence of ≥10% absolute decline in percentage of predicted FVC, ≥15% relative decline in 6MWT distance, lung transplantation, or death. FVC=pulmonary function test parameter that indicates the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It's measured by spirometry, which is a common breathing test to check lung function. 6MWT test is performed indoors on a flat, straight corridor with a hard surface at least 30 m in length. 6MWT measures the distance a participant is able to walk quickly on a flat, hard surface in a period of 6 minutes. 6MWT measure will be calculated as the simple difference between baseline distance walked over 6 minutes and week 52 distance walked over 6 minutes as measured in meters.
Cohorts 1 and 2: Time to First Acute Exacerbation of ILD, or Suspected Acute Exacerbation of ILD | From the start of study treatment until end of DBT (up to Week 52)
Cohorts 1 and 2: Change From Baseline in Quantitative Lung Fibrosis on High-Resolution Computed Tomography (HRCT) Scan of the Thorax | Baseline up to Week 52
  High-resolution computer tomography (HRCT) is a type of computed tomography (CT) with specific techniques to enhance image resolution. It is used in the diagnosis of various health problems, most commonly for lung disease. These images show cross sections (slices) through the lungs.
Cohorts 1 and 2: Percentage of Participants with Deaths | Up to Week 52
Cohort 2: Change From Baseline in Skin Sclerosis Assessed Using Modified Rodnan Skin Score (mRSS) | Baseline up to Week 52
  mRSS is a measure of skin thickness. Skin thickness will be assessed by the investigator by palpation across 17 different body sites and scored on a scale of 0 (normal) to 3 (severe skin thickening). The total score is the sum of the individual skin scores from all of these sites and ranges from 0 (normal) to 51 (severe thickening in all 17 areas) units. Higher scores indicate disease worsening.
Cohorts 1 and 2: Change From Baseline in Health-Related Quality of Life (HRQoL) Measured Using King's Brief Interstitial Lung Disease (K-BILD) Questionnaire | Baseline up to Week 52
  K-BILD is a questionnaire that assesses HRQoL in ILDs. It consists of 15 items grouped into psychological, breathlessness and activity, and chest symptom domains, each scored individually on a 7-point scale, with domain-level and total scores transformed 0-100, with higher scores indicating better quality of life. It uses a 2-week recall period.
Cohorts 1 and 2: Change From Baseline in Cough Measured Using Living with Pulmonary Fibrosis (L-PF) Symptoms Cough Domain Score | Baseline up to Week 52
  The L-PF symptoms module is a 23-item tool with domains capturing shortness of breath, cough, and energy symptoms using a 0-4 numeric response scale (NRS) response format and a 24-hour recall period. The cough scores ranges from 0 to 100 with higher scores indicating greater symptom burden/impairment.
Cohorts 1 and 2: Change From Baseline in Dyspnea Measured Using L-PF Symptoms Dyspnea Domain Score | Baseline up to Week 52
  The L-PF symptoms module is a 23-item tool with domains capturing shortness of breath, cough, and energy symptoms using a 0-4 NRS response format and a 24-hour recall period. L-PF Symptoms Dyspnea Domain score (dyspnea score) ranges from 0 to 100, with higher score indicating greater impairment.
Cohort 2: Change From Baseline in Pruritus Measured Using the Five-Dimension Itch Scale (5-D Itch) Total Score | Baseline up to Week 52
  The 5-D-Itch questionnaire that measures itch and its impact. It consists of 8 items organized into 5 domains (duration, degree, direction, disability, and distribution). Each domain is scored 1 to 5 with a total score ranging from 5 to 25 with higher scores indicating greater itch severity.
Cohorts 1, 2 and OLE Period: Number of Participants With Adverse Events (AEs) | Up to Week 52
Cohorts 1 and 2: Serum Concentration of Vixarelimab | Baseline up to Week 52
Cohorts 1 and 2: Number of Participants With Anti-Drug Antibodies (ADAs) to Vixarelimab | Baseline up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (114):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medicine Lung Institute, Phoenix, Arizona
  - Southern Arizona VA Health Care System NAVREF PPDS, Tucson, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - UCLA Rheumatology, Los Angeles, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - The Lundquist Institute for BioMedical Innovation at Harbor-UCLA Medical Cente, Torrance, California
  - Renstar Medical Research, Ocala, Florida
  - Coastal Pulmonary and Critical Care PLC, St. Petersburg, Florida
  - Weston Hospital, Weston, Florida
  - Piedmont Pulmonary and Sleep Medicine Buckhead, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - GenHarp Clinical Solutions, Evergreen Park, Illinois
  - Northwestern Medicine - Northwestern Medicine Glen, Glenview, Illinois
  - IU Health Ball Memorial Physicians Pulmonary and Critical Care Medicine, Muncie, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Hannibal Regional Healthcare System HRMG Hannibal, Hannibal, Missouri
  - Pulmonix LLC, Greensboro, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Baylor Scott and White Health - Advanced Lung Disease Specialists - Dallas, Dallas, Texas
  - IntraCare Health Center ? Prestige, Dallas, Texas
  - El Paso Pulmonary Association Elligo PPDS, El Paso, Texas
  - McGovern Medical School, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah - PPDS, Salt Lake City, Utah
- Argentina (11):
  - Centro Médico Dra de Salvo, Buenos Aires
  - Consultorios Médicos Dr. Doreski, Ciudad Autonoma Buenos Aires
  - Instituto Ave Pulmo, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
  - INSARES, Mendoza, Mendoza City
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
  - Instituto De Patologias Respiratorias, San Miguel de Tucumán
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
  - Centro de Investigaciones Reumatologicas, San Miguel de Tucumán
  - Instituto Del Buen Aire, Santa Fe
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Monash Health Monash Medical Centre, Clayton, Victoria
- Belgium (2):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - CHU de Liège, Liège
- Brazil (4):
  - L2 Ip - Instituto de Pesquisas Clinicas Ltda - ME, Brasília, Federal District
  - Hospital Brasilia, Brasília, Federal District
  - Hospital de Clinicas de Porto Alegre HCPA PPDS, Pôrto Alegre, Pará
  - Hospital Dia do Pulmao, Blumenau, Santa Catarina
- Canada (3):
  - Kelowna Allergy and Respiratory Health Clinic, Kelowna, British Columbia
  - Dynamic Drug Advancement Ltd., Ajax, Ontario
  - Dr Anil Dhar Professional Medicine Corporation, Windsor, Ontario
- Chile (3):
  - CEC SpA, Ñuñoa
  - Enroll SpA - PPDS, Providencia
  - Centro de Investigacion del Maule, Talca
- France (7):
  - Hopital Avicenne, Bobigny
  - Hopital Louis Pradel, Bron
  - Hopital Nord AP-HM, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hopital Pasteur 2, Nice
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - CHU de Reims, Reims
- Germany (3):
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Ruhrlandklinik, Essen
- Greece (2):
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
- Israel (9):
  - Barzilai Medical Center, Ashkelon
  - Shamir Medical Center Assaf Harofeh, Beer Jacob
  - Rambam Medical Center, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (9):
  - Azienda Ospedaliera Universitaria Senese, Siena, Abruzzo
  - Presidio Ospedaliero GB Morgagni L Pierantoni, Forlì, Emilia-Romagna
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Ospedale S. Giuseppe Multimedica, Milan, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliera Universitaria "Policlinico - Vittorio Emanuele" (Presidio Gaspare Rodolico), Catania, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona, The Marches
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
- Mexico (3):
  - CICUM San Miguel, Americana, Jalisco
  - Bioclinica - Centro Integral En Reumatologia Sociedad Anónima de Capital Variable - PPDS, Guadalajara, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- Poland (4):
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów
  - PULMAG Grzegorz Gasior Marzena Kociolek Spolka Cywilna, Sosnowiec
  - Wojskowy Instytut Medyczny Panstwowy Instytut Badawczy, Warsaw
- South Africa (3):
  - Dr JM Engelbrecht Trial site, Cape Town
  - University of Cape Town Lung Institute UCTLI, Cape Town
  - St Augustines Hospital, Durban
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
- Spain (9):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - CHUS H Clinico U de Santiago, Santiago de Compostela, LA Coruna
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca
- Taiwan (3):
  - Far East Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing